CLINICAL TRIAL: NCT01170728
Title: Virtue® Male Sling Fixation Study
Status: Terminated | Type: Observational
Why Stopped: The study has been terminated due to lack of subject enrollment.
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP008SU
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Male Sling; Fixation; Stress Urinary Incontinence; Urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Virtue® Male Sling: Device: Coloplast Virtue® Male Sling
  Interventions: Device: Coloplast Virtue® Male Sling

INTERVENTIONS:
Device: Coloplast Virtue® Male Sling — The Virtue Male sling is a class II single use implantable sub-urethral, permanent, non-absorbable, support sling indicated for the surgical treatment of male stress urinary incontinence (SUI) resulting from intrinsic sphincter deficiency (ISD). The device consists of a knitted monofilament polypropylene mesh which provides surface area for supporting the bulbous urethra. The four arms are covered with polyethylene sleeves with braided polyester sutures attached at the end of the mesh arms providing proper attachment to the introducer for positioning of the sling. The single use introducer allows for implanting both the trans-obturator arms and pre-pubic arms of the mesh sling.

SUMMARY:
This study is a multi-center study that will assess the efficacy and safety of suture fixation of the Virtue® Male Sling.

ELIGIBILITY:
Inclusion Criteria:

* Male subject at least 18 years of age with an estimated life expectancy of of more than 5 years
* The subject has confirmed stress urinary incontinence (SUI) through medical history , urodynamics, and/or physical exam for at least 6 months
* The subject has completed post-void residual per protocol within 6 weeks prior to implant
* The subject has completed cystoscopy as per protocol within 12 months prior to implant
* The subject has intrinsic sphincter deficiency due to one of the following: post-transurethral resection of the prostate (TURP), simple open prostatectomy, or radical prostatectomy completed at least 6 months prior to implantation date
* The subject has failed at least two non-invasive therapies, eg. pelvic/Kegel exercises, behavioral modification or biofeedback for at least 6 months
* The subject is willing to have the Virtue® Male Sling implanted
* The subject is able and willing to complete all follow-up visits and procedures indicated in the protocol
* The subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the local ethics committee of the respective site

Exclusion Criteria:

* The subject is unable or unwilling to sign the informed consent form (ICF)and/or comply with all follow-up requirements according to the study protocol
* The subject has an active urinary tract infection or active skin infection in region of surgery
* The subject has serious bleeding disorders
* The subject has incontinence due to neurogenic causes defined as multiple sclerosis, spinal cord/brain injury, cerebrovascular accident (CVA), detrusor-external sphincter dyssynergia, Parkinson's disease, or similar condition
* The subject had a previous implant to treat stress urinary incontinence
* The subject has undergone radiation, cryosurgery, or brachy therapy to treat prostate or other pelvic cancer within 6 months
* The subject is likely to undergo radiation therapy within the next 6 months
* The subject has active urethral or bladder neck stricture disease requiring continued treatment
* The subject has urge predominant incontinence
* The subject has an atonic bladder or a postvoid residual (PVR) greater than or equal to 150 milliliters (mL)
* The subject has a condition or disorder likely to require future transurethral procedure
* The subject is enrolled in a concurrent clinical study of any treatment (drug or device) that could affect continence function without sponsor's approval
* The subject is deemed unfit for male sling implantation or participation in a research protocol as determined by attending physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects satisfying inclusion and exclusion criteria were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Improvement of incontinence | 3 months post implant
Safety of the device characterized by reported adverse events | 3 months

SECONDARY OUTCOMES:
To characterize incontinence severity at various time points | 24 months
To evaluate patient quality of life at specified time points | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig Comiter, MD, Study Chair — Stanford University
Locations (10):
- United States (10):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Kaiser Permanente, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Winter Park Urology, Orlando, Florida
  - Midtown Urology, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - NYU Urology Associates, New York, New York
  - McKay Urology, Charlotte, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates of North Texas, Arlington, Texas